CLINICAL TRIAL: NCT01286454
Title: An Open-Label, Single-Dose, Randomized, Cross-Over Study To Estimate The Bioavailability And Food Effect Of 4 Mg Fesoterodine Extended Release Beads-In-Capsule Formulations Compared To Commercial Tablet Formulation In Healthy Volunteers
Brief Title: This Is A Study Of Bioavailability And Food Effect For Fesoterodine.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A0221068
Record Dates: First submitted 2010-12-03; First posted 2011-01-31 (Estimated); Results first posted 2012-01-09 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Overactive Bladder (OAB) With Symptoms of Frequency, Urgency, and Urgency
Keywords: BIOAVAILABILITY; FOOD EFFECT
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- A (Experimental): 4 mg fesoterodine IR beads in capsule under fasting condition
  Interventions: Drug: fesoterodine
- B (Experimental): 4 mg fesoterodine 10% coated ER beads in capsule under fasting condition
  Interventions: Drug: fesoterodine
- C (Experimental): 4 mg fesoterodine 15% coated ER beads in capsule under fasting condition.
  Interventions: Drug: fesoterodine
- D (Experimental): 4 mg fesoterodine 20% coated ER beads in capsule under fasting condition.
  Interventions: Drug: fesoterodine
- E (Experimental): 4 mg fesoterodine ER tablets under fasting condition.
  Interventions: Drug: fesoterodine
- F (Experimental): 4 mg fesoterodine TBD % coated ER beads in capsule under fed condition.
  Interventions: Drug: fesoterodine

INTERVENTIONS:
Drug: fesoterodine — single dose of beads in capsule
  Arms: A
Drug: fesoterodine — single dose of beads in capsule
  Arms: B
Drug: fesoterodine — single dose of beads in capsule
  Arms: C
Drug: fesoterodine — single dose of beads in capsule
  Arms: D
Drug: fesoterodine — single dose of tablet
  Arms: E
Drug: fesoterodine — single dose of beads in capsule
  Arms: F

SUMMARY:
This Is A Study Of Bioavailability And Food Effect For Fesoterodine.

DETAILED DESCRIPTION:
To estimate the bioavailability of three different 4 mg fesoterodine ER beads-incapsule formulations compared to 4 mg fesoterodine marketed ER tablets under fasting and fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years

Exclusion Criteria:

* Evidence or history of clinically significant disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221068&StudyName=This%20Is%20A%20Study%20Of%20Bioavailability%20And%20Food%20Effect%20For%20Fesoterodine.

RESULTS

PARTICIPANT FLOW:
Groups:
- Fesoterodine 4mg IR, 10% ER, ER Tablet, 15% ER, 20% ER: Single oral dose of fesoterodine 4 milligram (mg) immediate release (IR) beads-in-capsule (BIC) under fasted condition in first intervention period; followed by single oral dose of fesoterodine 4 mg 10% coated extended release (ER) BIC under fasted condition in second intervention period; then single oral dose of fesoterodine 4 mg ER tablet under fasted condition in third intervention period; then single oral dose of fesoterodine 4 mg 15% coated ER-BIC under fasted condition in fourth intervention period; and single oral dose of fesoterodine 4 mg 20% coated ER-BIC under fasted condition in fifth intervention period. A washout period of at least 3 days between intervention periods was maintained.
- Fesoterodine 4mg 10% ER, 15% ER, IR, 20% ER, ER Tablet: Single oral dose of fesoterodine 4 mg 10% coated ER-BIC under fasted condition in first intervention period; followed by single oral dose of fesoterodine 4 mg 15% coated ER-BIC under fasted condition in second intervention period; then single oral dose of fesoterodine 4 mg IR-BIC under fasted condition in third intervention period; then single oral dose of fesoterodine 4 mg 20% coated ER-BIC under fasted condition in forth intervention period; and single oral dose of fesoterodine 4 mg ER tablet under fasted condition in fifth intervention period. A washout period of at least 3 days between intervention periods was maintained.
- Fesoterodine 4mg 15% ER, 20% ER, 10% ER, ER Tablet, IR: Single oral dose of fesoterodine 4 mg 15% coated ER-BIC under fasted condition in first intervention period; followed by single oral dose of fesoterodine 4 mg 20% coated ER-BIC under fasted condition in second intervention period; then single oral dose of fesoterodine 4 mg 10% coated ER-BIC under fasted condition in third intervention period; then single oral dose of fesoterodine 4 mg ER tablet under fasted condition in fourth intervention period; and single oral dose of fesoterodine 4 mg IR-BIC under fasted condition in fifth intervention period. A washout period of at least 3 days between intervention periods was maintained.
- Fesoterodine 4mg 20% ER, ER Tablet, 15% ER, IR, 10% ER: Single oral dose of fesoterodine 4 mg 20% coated ER-BIC under fasted condition in first intervention period; followed by single oral dose of fesoterodine 4 mg ER tablet under fasted condition in second intervention period; then single oral dose of fesoterodine 4 mg 15% coated ER-BIC under fasted condition in third intervention period; then single oral dose of fesoterodine 4 mg IR-BIC under fasted condition in fourth intervention period; and single oral dose of fesoterodine 4 mg 10% coated ER-BIC under fasted condition in fifth intervention period. A washout period of at least 3 days between intervention periods was maintained.
- Fesoterodine 4mg ER Tablet, IR, 20% ER, 10% ER, 15% ER: Single oral dose of fesoterodine 4 mg ER tablet under fasted condition in first intervention period; followed by single oral dose of fesoterodine 4 mg IR-BIC under fasted condition in second intervention period; then single oral dose of fesoterodine 4 mg 20% coated ER-BIC under fasted condition in third intervention period; then single oral dose of fesoterodine 4 mg 10% coated ER-BIC under fasted condition in fourth intervention period; and single oral dose of fesoterodine 4 mg 15% coated ER-BIC under fasted condition in fifth intervention period. A washout period of at least 3 days between intervention periods was maintained.
- Fesoterodine 4mg IR, ER Tablet, 10% ER, 20% ER, 15% ER: Single oral dose of fesoterodine 4 mg IR-BIC under fasted condition in first intervention period; followed by single oral dose of fesoterodine 4 mg ER tablet under fasted condition in second intervention period; then single oral dose of fesoterodine 4 mg 10% coated ER-BIC under fasted condition in third intervention period; then single oral dose of fesoterodine 4 mg 20% coated ER-BIC under fasted condition in fourth intervention period; and single oral dose of fesoterodine 4 mg 15% coated ER-BIC under fasted condition in fifth intervention period. A washout period of at least 3 days between intervention periods was maintained.
- Fesoterodine 4mg 10% ER, IR, 15% ER, ER Tablet, 20% ER: Single oral dose of fesoterodine 4 mg 10% coated ER-BIC under fasted condition in first intervention period; followed by single oral dose of fesoterodine 4 mg IR-BIC under fasted condition in second intervention period; then single oral dose of fesoterodine 4 mg 15% coated ER-BIC under fasted condition in third intervention period; then single oral dose of fesoterodine 4 mg ER tablet under fasted condition in fourth intervention period; and single oral dose of fesoterodine 4 mg 20% coated ER-BIC under fasted condition in fifth intervention period. A washout period of at least 3 days between intervention periods was maintained.
- Fesoterodine 4mg 15% ER, 10% ER, 20% ER, IR, ER Tablet: Single oral dose of fesoterodine 4 mg 15% coated ER-BIC under fasted condition in first intervention period; followed by single oral dose of fesoterodine 4 mg 10% coated ER-BIC under fasted condition in second intervention period; then single oral dose of fesoterodine 4 mg 20% coated ER-BIC under fasted condition in third intervention period; then single oral dose of fesoterodine 4 mg IR-BIC under fasted condition in fourth intervention period; and single oral dose of fesoterodine 4 mg ER tablet under fasted condition in fifth intervention period. A washout period of at least 3 days between intervention periods was maintained.
- Fesoterodine 4mg 20% ER, 15% ER, ER Tablet, 10% ER, IR: Single oral dose of fesoterodine 4 mg 20% coated ER-BIC under fasted condition in first intervention period; followed by single oral dose of fesoterodine 4 mg 15% coated ER-BIC under fasted condition in second intervention period; then single oral dose of fesoterodine 4 mg ER tablet under fasted condition in third intervention period; then single oral dose of fesoterodine 4 mg 10% coated ER-BIC under fasted condition in fourth intervention period; and single oral dose of fesoterodine 4 mg IR-BIC under fasted condition in fifth intervention period. A washout period of at least 3 days between intervention periods was maintained.
- Fesoterodine 4mg ER Tablet, 20% ER, IR, 15% ER, 10% ER: Single oral dose of fesoterodine 4 mg ER tablet under fasted condition in first intervention period; followed by single oral dose of fesoterodine 4 mg 20% coated ER-BIC under fasted condition in second intervention period; then single oral dose of fesoterodine 4 mg IR-BIC under fasted condition in third intervention period; then single oral dose of fesoterodine 4 mg 15% coated ER-BIC under fasted condition in fourth intervention period; and single oral dose of fesoterodine 4 mg 10% coated ER-BIC under fasted condition in fifth intervention period. A washout period of at least 3 days between intervention periods was maintained.
- Fesoterodine 4 mg 10% ER Fed: Single oral dose of fesoterodine 4 mg 10% coated ER-BIC under fed condition in sixth intervention period. A washout period of approximately 2 weeks was maintained between fifth and sixth intervention period.
Period: Part I- First Intervention Period
Arm/Group | Fesoterodine 4mg IR, 10% ER, ER Tablet, 15% ER, 20% ER | Fesoterodine 4mg 10% ER, 15% ER, IR, 20% ER, ER Tablet | Fesoterodine 4mg 15% ER, 20% ER, 10% ER, ER Tablet, IR | Fesoterodine 4mg 20% ER, ER Tablet, 15% ER, IR, 10% ER | Fesoterodine 4mg ER Tablet, IR, 20% ER, 10% ER, 15% ER | Fesoterodine 4mg IR, ER Tablet, 10% ER, 20% ER, 15% ER | Fesoterodine 4mg 10% ER, IR, 15% ER, ER Tablet, 20% ER | Fesoterodine 4mg 15% ER, 10% ER, 20% ER, IR, ER Tablet | Fesoterodine 4mg 20% ER, 15% ER, ER Tablet, 10% ER, IR | Fesoterodine 4mg ER Tablet, 20% ER, IR, 15% ER, 10% ER | Fesoterodine 4 mg 10% ER Fed
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (At Least 3 Days)
Arm/Group | Fesoterodine 4mg IR, 10% ER, ER Tablet, 15% ER, 20% ER | Fesoterodine 4mg 10% ER, 15% ER, IR, 20% ER, ER Tablet | Fesoterodine 4mg 15% ER, 20% ER, 10% ER, ER Tablet, IR | Fesoterodine 4mg 20% ER, ER Tablet, 15% ER, IR, 10% ER | Fesoterodine 4mg ER Tablet, IR, 20% ER, 10% ER, 15% ER | Fesoterodine 4mg IR, ER Tablet, 10% ER, 20% ER, 15% ER | Fesoterodine 4mg 10% ER, IR, 15% ER, ER Tablet, 20% ER | Fesoterodine 4mg 15% ER, 10% ER, 20% ER, IR, ER Tablet | Fesoterodine 4mg 20% ER, 15% ER, ER Tablet, 10% ER, IR | Fesoterodine 4mg ER Tablet, 20% ER, IR, 15% ER, 10% ER | Fesoterodine 4 mg 10% ER Fed
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention Period
Arm/Group | Fesoterodine 4mg IR, 10% ER, ER Tablet, 15% ER, 20% ER | Fesoterodine 4mg 10% ER, 15% ER, IR, 20% ER, ER Tablet | Fesoterodine 4mg 15% ER, 20% ER, 10% ER, ER Tablet, IR | Fesoterodine 4mg 20% ER, ER Tablet, 15% ER, IR, 10% ER | Fesoterodine 4mg ER Tablet, IR, 20% ER, 10% ER, 15% ER | Fesoterodine 4mg IR, ER Tablet, 10% ER, 20% ER, 15% ER | Fesoterodine 4mg 10% ER, IR, 15% ER, ER Tablet, 20% ER | Fesoterodine 4mg 15% ER, 10% ER, 20% ER, IR, ER Tablet | Fesoterodine 4mg 20% ER, 15% ER, ER Tablet, 10% ER, IR | Fesoterodine 4mg ER Tablet, 20% ER, IR, 15% ER, 10% ER | Fesoterodine 4 mg 10% ER Fed
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (At Least 3 Days)
Arm/Group | Fesoterodine 4mg IR, 10% ER, ER Tablet, 15% ER, 20% ER | Fesoterodine 4mg 10% ER, 15% ER, IR, 20% ER, ER Tablet | Fesoterodine 4mg 15% ER, 20% ER, 10% ER, ER Tablet, IR | Fesoterodine 4mg 20% ER, ER Tablet, 15% ER, IR, 10% ER | Fesoterodine 4mg ER Tablet, IR, 20% ER, 10% ER, 15% ER | Fesoterodine 4mg IR, ER Tablet, 10% ER, 20% ER, 15% ER | Fesoterodine 4mg 10% ER, IR, 15% ER, ER Tablet, 20% ER | Fesoterodine 4mg 15% ER, 10% ER, 20% ER, IR, ER Tablet | Fesoterodine 4mg 20% ER, 15% ER, ER Tablet, 10% ER, IR | Fesoterodine 4mg ER Tablet, 20% ER, IR, 15% ER, 10% ER | Fesoterodine 4 mg 10% ER Fed
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention Period
Arm/Group | Fesoterodine 4mg IR, 10% ER, ER Tablet, 15% ER, 20% ER | Fesoterodine 4mg 10% ER, 15% ER, IR, 20% ER, ER Tablet | Fesoterodine 4mg 15% ER, 20% ER, 10% ER, ER Tablet, IR | Fesoterodine 4mg 20% ER, ER Tablet, 15% ER, IR, 10% ER | Fesoterodine 4mg ER Tablet, IR, 20% ER, 10% ER, 15% ER | Fesoterodine 4mg IR, ER Tablet, 10% ER, 20% ER, 15% ER | Fesoterodine 4mg 10% ER, IR, 15% ER, ER Tablet, 20% ER | Fesoterodine 4mg 15% ER, 10% ER, 20% ER, IR, ER Tablet | Fesoterodine 4mg 20% ER, 15% ER, ER Tablet, 10% ER, IR | Fesoterodine 4mg ER Tablet, 20% ER, IR, 15% ER, 10% ER | Fesoterodine 4 mg 10% ER Fed
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (At Least 3 Days)
Arm/Group | Fesoterodine 4mg IR, 10% ER, ER Tablet, 15% ER, 20% ER | Fesoterodine 4mg 10% ER, 15% ER, IR, 20% ER, ER Tablet | Fesoterodine 4mg 15% ER, 20% ER, 10% ER, ER Tablet, IR | Fesoterodine 4mg 20% ER, ER Tablet, 15% ER, IR, 10% ER | Fesoterodine 4mg ER Tablet, IR, 20% ER, 10% ER, 15% ER | Fesoterodine 4mg IR, ER Tablet, 10% ER, 20% ER, 15% ER | Fesoterodine 4mg 10% ER, IR, 15% ER, ER Tablet, 20% ER | Fesoterodine 4mg 15% ER, 10% ER, 20% ER, IR, ER Tablet | Fesoterodine 4mg 20% ER, 15% ER, ER Tablet, 10% ER, IR | Fesoterodine 4mg ER Tablet, 20% ER, IR, 15% ER, 10% ER | Fesoterodine 4 mg 10% ER Fed
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Fourth Intervention Period
Arm/Group | Fesoterodine 4mg IR, 10% ER, ER Tablet, 15% ER, 20% ER | Fesoterodine 4mg 10% ER, 15% ER, IR, 20% ER, ER Tablet | Fesoterodine 4mg 15% ER, 20% ER, 10% ER, ER Tablet, IR | Fesoterodine 4mg 20% ER, ER Tablet, 15% ER, IR, 10% ER | Fesoterodine 4mg ER Tablet, IR, 20% ER, 10% ER, 15% ER | Fesoterodine 4mg IR, ER Tablet, 10% ER, 20% ER, 15% ER | Fesoterodine 4mg 10% ER, IR, 15% ER, ER Tablet, 20% ER | Fesoterodine 4mg 15% ER, 10% ER, 20% ER, IR, ER Tablet | Fesoterodine 4mg 20% ER, 15% ER, ER Tablet, 10% ER, IR | Fesoterodine 4mg ER Tablet, 20% ER, IR, 15% ER, 10% ER | Fesoterodine 4 mg 10% ER Fed
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (At Least 3 Days)
Arm/Group | Fesoterodine 4mg IR, 10% ER, ER Tablet, 15% ER, 20% ER | Fesoterodine 4mg 10% ER, 15% ER, IR, 20% ER, ER Tablet | Fesoterodine 4mg 15% ER, 20% ER, 10% ER, ER Tablet, IR | Fesoterodine 4mg 20% ER, ER Tablet, 15% ER, IR, 10% ER | Fesoterodine 4mg ER Tablet, IR, 20% ER, 10% ER, 15% ER | Fesoterodine 4mg IR, ER Tablet, 10% ER, 20% ER, 15% ER | Fesoterodine 4mg 10% ER, IR, 15% ER, ER Tablet, 20% ER | Fesoterodine 4mg 15% ER, 10% ER, 20% ER, IR, ER Tablet | Fesoterodine 4mg 20% ER, 15% ER, ER Tablet, 10% ER, IR | Fesoterodine 4mg ER Tablet, 20% ER, IR, 15% ER, 10% ER | Fesoterodine 4 mg 10% ER Fed
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Fifth Intervention Period
Arm/Group | Fesoterodine 4mg IR, 10% ER, ER Tablet, 15% ER, 20% ER | Fesoterodine 4mg 10% ER, 15% ER, IR, 20% ER, ER Tablet | Fesoterodine 4mg 15% ER, 20% ER, 10% ER, ER Tablet, IR | Fesoterodine 4mg 20% ER, ER Tablet, 15% ER, IR, 10% ER | Fesoterodine 4mg ER Tablet, IR, 20% ER, 10% ER, 15% ER | Fesoterodine 4mg IR, ER Tablet, 10% ER, 20% ER, 15% ER | Fesoterodine 4mg 10% ER, IR, 15% ER, ER Tablet, 20% ER | Fesoterodine 4mg 15% ER, 10% ER, 20% ER, IR, ER Tablet | Fesoterodine 4mg 20% ER, 15% ER, ER Tablet, 10% ER, IR | Fesoterodine 4mg ER Tablet, 20% ER, IR, 15% ER, 10% ER | Fesoterodine 4 mg 10% ER Fed
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (Approximately 2 Weeks)
Arm/Group | Fesoterodine 4mg IR, 10% ER, ER Tablet, 15% ER, 20% ER | Fesoterodine 4mg 10% ER, 15% ER, IR, 20% ER, ER Tablet | Fesoterodine 4mg 15% ER, 20% ER, 10% ER, ER Tablet, IR | Fesoterodine 4mg 20% ER, ER Tablet, 15% ER, IR, 10% ER | Fesoterodine 4mg ER Tablet, IR, 20% ER, 10% ER, 15% ER | Fesoterodine 4mg IR, ER Tablet, 10% ER, 20% ER, 15% ER | Fesoterodine 4mg 10% ER, IR, 15% ER, ER Tablet, 20% ER | Fesoterodine 4mg 15% ER, 10% ER, 20% ER, IR, ER Tablet | Fesoterodine 4mg 20% ER, 15% ER, ER Tablet, 10% ER, IR | Fesoterodine 4mg ER Tablet, 20% ER, IR, 15% ER, 10% ER | Fesoterodine 4 mg 10% ER Fed
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part II- Sixth Intervention Period
Arm/Group | Fesoterodine 4mg IR, 10% ER, ER Tablet, 15% ER, 20% ER | Fesoterodine 4mg 10% ER, 15% ER, IR, 20% ER, ER Tablet | Fesoterodine 4mg 15% ER, 20% ER, 10% ER, ER Tablet, IR | Fesoterodine 4mg 20% ER, ER Tablet, 15% ER, IR, 10% ER | Fesoterodine 4mg ER Tablet, IR, 20% ER, 10% ER, 15% ER | Fesoterodine 4mg IR, ER Tablet, 10% ER, 20% ER, 15% ER | Fesoterodine 4mg 10% ER, IR, 15% ER, ER Tablet, 20% ER | Fesoterodine 4mg 15% ER, 10% ER, 20% ER, IR, ER Tablet | Fesoterodine 4mg 20% ER, 15% ER, ER Tablet, 10% ER, IR | Fesoterodine 4mg ER Tablet, 20% ER, IR, 15% ER, 10% ER | Fesoterodine 4 mg 10% ER Fed
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive fesoterodine 4 mg IR-BIC fasted first, 10% ER-BIC fasted first, 15% ER-BIC fasted first, 20% ER-BIC fasted first and ER tablets fasted first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 39.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] for Fesoterodine Metabolite (5-hydroxymethyltolterodine [5-HMT])
Description: AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 30, 36 and 48 hours (hrs) post dose
Population: Pharmacokinetic (PK) parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period. Here, the N (number of participants analyzed) is signifying the number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Fesoterodine 4 mg IR-BIC Fasted: Single oral dose of fesoterodine 4 mg IR-BIC under fasted condition in either of the first to fifth intervention periods.
- Fesoterodine 4 mg 10% ER-BIC Fasted: Single oral dose of fesoterodine 4 mg 10% coated ER-BIC under fasted condition in either of the first to fifth intervention periods.
- Fesoterodine 4 mg 15% ER-BIC Fasted: Single oral dose of fesoterodine 4 mg 15% coated ER-BIC under fasted condition in either of the first to fifth intervention periods.
- Fesoterodine 4 mg 20% ER-BIC Fasted: Single oral dose of fesoterodine 4 mg 20% coated ER-BIC under fasted condition in either of the first to fifth intervention periods.
- Fesoterodine 4 mg ER Tablet Fasted: Single oral dose of fesoterodine 4 mg ER Tablet under fasted condition in either of the first to fifth intervention periods.
- Fesoterodine 4 mg 10% ER-BIC Fed: Single oral dose of fesoterodine 4 mg 10% coated ER-BIC under fed condition in the sixth intervention period.
Arm/Group | Fesoterodine 4 mg IR-BIC Fasted | Fesoterodine 4 mg 10% ER-BIC Fasted | Fesoterodine 4 mg 15% ER-BIC Fasted | Fesoterodine 4 mg 20% ER-BIC Fasted | Fesoterodine 4 mg ER Tablet Fasted | Fesoterodine 4 mg 10% ER-BIC Fed
Number analyzed (Participants) | 20 | 20 | 16 | 4 | 20 | 20
ng*hr/mL | 30.48 (11.77) | 28.24 (10.35) | 19.64 (7.58) | NA (NA) — Parameter was missing for more than 50 percent of the participants. | 27.40 (10.06) | 32.07 (13.24)
Statistical Analysis 1: Comparison: Fesoterodine 4 mg IR-BIC Fasted vs Fesoterodine 4 mg ER Tablet Fasted; Natural log transformed AUC (0 - ∞) of 5-HMT was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% confidence intervals (CIs) for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. Fesoterodine 4 mg ER Tablet Fasted was reference and Fesoterodine 4 mg IR-BIC Fasted was test; Test type: Superiority or Other; Ratio of Adjusted Means = 111.23, 90% CI 2-sided [102.69 to 120.47]
Statistical Analysis 2: Comparison: Fesoterodine 4 mg 10% ER-BIC Fasted vs Fesoterodine 4 mg ER Tablet Fasted; Natural log transformed AUC (0 - ∞) of 5-HMT was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. Fesoterodine 4 mg ER Tablet Fasted was reference and Fesoterodine 4 mg 10% ER-BIC Fasted was test; Test type: Superiority or Other; Ratio of Adjusted Means = 103.07, 90% CI 2-sided [95.16 to 111.64]
Statistical Analysis 3: Comparison: Fesoterodine 4 mg 15% ER-BIC Fasted vs Fesoterodine 4 mg ER Tablet Fasted; Natural log transformed AUC (0 - ∞) of 5-HMT was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. Fesoterodine 4 mg ER Tablet Fasted was reference and Fesoterodine 4 mg 15% ER-BIC Fasted was test; Test type: Superiority or Other; Ratio of Adjusted Means = 70.36, 90% CI 2-sided [64.52 to 76.74]
Statistical Analysis 4: Comparison: Fesoterodine 4 mg 10% ER-BIC Fasted vs Fesoterodine 4 mg 10% ER-BIC Fed; Natural log transformed AUC (0 - ∞) of 5-HMT was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. Fesoterodine 4 mg 10% ER-BIC Fasted was reference and Fesoterodine 4 mg 10% ER-BIC Fed was test; Test type: Superiority or Other; Ratio of Adjusted Means = 113.55, 90% CI 2-sided [105.91 to 121.74]

2. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for Fesoterodine Metabolite (5-HMT)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast) of 5-HMT.
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 30, 36 and 48 hrs post dose
Population: PK parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Fesoterodine 4 mg IR-BIC Fasted | Fesoterodine 4 mg 10% ER-BIC Fasted | Fesoterodine 4 mg 15% ER-BIC Fasted | Fesoterodine 4 mg 20% ER-BIC Fasted | Fesoterodine 4 mg ER Tablet Fasted | Fesoterodine 4 mg 10% ER-BIC Fed
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
ng*hr/mL | 30.23 (11.79) | 27.79 (10.21) | 17.92 (6.95) | 7.59 (3.57) | 26.80 (10.07) | 31.88 (13.24)
Statistical Analysis 1: Comparison: Fesoterodine 4 mg IR-BIC Fasted vs Fesoterodine 4 mg ER Tablet Fasted; Natural log transformed AUClast of 5-HMT was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. Fesoterodine 4 mg ER Tablet Fasted was reference and Fesoterodine 4 mg IR-BIC Fasted was test; Test type: Superiority or Other; Ratio of Adjusted Means = 112.80, 90% CI 2-sided [103.85 to 122.52]
Statistical Analysis 2: Comparison: Fesoterodine 4 mg 10% ER-BIC Fasted vs Fesoterodine 4 mg ER Tablet Fasted; Natural log transformed AUClast of 5-HMT was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. Fesoterodine 4 mg ER Tablet Fasted was reference and Fesoterodine 4 mg 10% ER-BIC Fasted was test; Test type: Superiority or Other; Ratio of Adjusted Means = 103.71, 90% CI 2-sided [95.48 to 112.65]
Statistical Analysis 3: Comparison: Fesoterodine 4 mg 15% ER-BIC Fasted vs Fesoterodine 4 mg ER Tablet Fasted; Natural log transformed AUClast of 5-HMT was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. Fesoterodine 4 mg ER Tablet Fasted was reference and Fesoterodine 4 mg 15% ER-BIC Fasted was test; Test type: Superiority or Other; Ratio of Adjusted Means = 66.87, 90% CI 2-sided [61.56 to 72.63]
Statistical Analysis 4: Comparison: Fesoterodine 4 mg 20% ER-BIC Fasted vs Fesoterodine 4 mg ER Tablet Fasted; Natural log transformed AUClast of 5-HMT was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. Fesoterodine 4 mg ER Tablet Fasted was reference and Fesoterodine 4 mg 20% ER-BIC Fasted was test; Test type: Superiority or Other; Ratio of Adjusted Means = 28.34, 90% CI 2-sided [26.09 to 30.78]
Statistical Analysis 5: Comparison: Fesoterodine 4 mg 10% ER-BIC Fasted vs Fesoterodine 4 mg 10% ER-BIC Fed; Natural log transformed AUClast of 5-HMT was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. Fesoterodine 4 mg 10% ER-BIC Fasted was reference and Fesoterodine 4 mg 10% ER-BIC Fed was test; Test type: Superiority or Other; Ratio of Adjusted Means = 114.70, 90% CI 2-sided [106.99 to 122.97]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for Fesoterodine Metabolite (5-HMT)
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 30, 36 and 48 hrs post dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Fesoterodine 4 mg IR-BIC Fasted | Fesoterodine 4 mg 10% ER-BIC Fasted | Fesoterodine 4 mg 15% ER-BIC Fasted | Fesoterodine 4 mg 20% ER-BIC Fasted | Fesoterodine 4 mg ER Tablet Fasted | Fesoterodine 4 mg 10% ER-BIC Fed
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
ng/mL | 5.830 (2.729) | 3.030 (1.068) | 1.092 (0.496) | 0.323 (0.183) | 2.247 (1.000) | 5.183 (1.919)
Statistical Analysis 1: Comparison: Fesoterodine 4 mg IR-BIC Fasted vs Fesoterodine 4 mg ER Tablet Fasted; Natural log transformed Cmax of 5-HMT was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. Fesoterodine 4 mg ER Tablet Fasted was reference and Fesoterodine 4 mg IR-BIC Fasted was test; Test type: Superiority or Other; Ratio of Adjusted Means = 259.40, 90% CI 2-sided [231.48 to 290.70]
Statistical Analysis 2: Comparison: Fesoterodine 4 mg 10% ER-BIC Fasted vs Fesoterodine 4 mg ER Tablet Fasted; Natural log transformed Cmax of 5-HMT was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. Fesoterodine 4 mg ER Tablet Fasted was reference and Fesoterodine 4 mg 10% ER-BIC Fasted was test; Test type: Superiority or Other; Ratio of Adjusted Means = 134.83, 90% CI 2-sided [120.31 to 151.09]
Statistical Analysis 3: Comparison: Fesoterodine 4 mg 15% ER-BIC Fasted vs Fesoterodine 4 mg ER Tablet Fasted; Natural log transformed Cmax of 5-HMT was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. Fesoterodine 4 mg ER Tablet Fasted was reference and Fesoterodine 4 mg 15% ER-BIC Fasted was test; Test type: Superiority or Other; Ratio of Adjusted Means = 48.58, 90% CI 2-sided [43.35 to 54.44]
Statistical Analysis 4: Comparison: Fesoterodine 4 mg 20% ER-BIC Fasted vs Fesoterodine 4 mg ER Tablet Fasted; Natural log transformed Cmax of 5-HMT was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. Fesoterodine 4 mg ER Tablet Fasted was reference and Fesoterodine 4 mg 20% ER-BIC Fasted was test; Test type: Superiority or Other; Ratio of Adjusted Means = 14.38, 90% CI 2-sided [12.83 to 16.11]
Statistical Analysis 5: Comparison: Fesoterodine 4 mg 10% ER-BIC Fasted vs Fesoterodine 4 mg 10% ER-BIC Fed; Natural log transformed Cmax of 5-HMT was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. Fesoterodine 4 mg 10% ER-BIC Fasted was reference and Fesoterodine 4 mg 10% ER-BIC Fed was test; Test type: Superiority or Other; Ratio of Adjusted Means = 171.06, 90% CI 2-sided [115.82 to 187.78]

4. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for Fesoterodine Metabolite (5-HMT)
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 30, 36 and 48 hrs post dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Fesoterodine 4 mg IR-BIC Fasted | Fesoterodine 4 mg 10% ER-BIC Fasted | Fesoterodine 4 mg 15% ER-BIC Fasted | Fesoterodine 4 mg 20% ER-BIC Fasted | Fesoterodine 4 mg ER Tablet Fasted | Fesoterodine 4 mg 10% ER-BIC Fed
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
hr | 1.0 [0.5 to 5.0] | 6.0 [5.0 to 8.0] | 6.0 [5.0 to 10.0] | 8.0 [5.0 to 24.0] | 5.0 [2.0 to 6.0] | 4.0 [3.0 to 6.0]

5. Secondary Outcome: Plasma Decay Half Life (t1/2) for Fesoterodine Metabolite (5-HMT)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 30, 36 and 48 hrs post dose
Population: PK parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period. Here, the N (number of participants analyzed) is signifying the number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Fesoterodine 4 mg IR-BIC Fasted | Fesoterodine 4 mg 10% ER-BIC Fasted | Fesoterodine 4 mg 15% ER-BIC Fasted | Fesoterodine 4 mg 20% ER-BIC Fasted | Fesoterodine 4 mg ER Tablet Fasted | Fesoterodine 4 mg 10% ER-BIC Fed
Number analyzed (Participants) | 20 | 20 | 16 | 4 | 20 | 20
hr | 5.56 (1.70) | 7.22 (1.68) | 10.89 (4.45) | NA (NA) — Parameter was missing for more than 50 percent of the participants. | 7.54 (2.49) | 4.59 (0.76)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Fesoterodine 4 mg IR-BIC Fasted | Fesoterodine 4 mg 10% ER-BIC Fasted | Fesoterodine 4 mg 15% ER-BIC Fasted | Fesoterodine 4 mg 20% ER-BIC Fasted | Fesoterodine 4 mg ER Tablet Fasted | Fesoterodine 4 mg 10% ER-BIC Fed
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 7/20 | 4/20 | 6/20 | 0/20 | 4/20 | 6/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine 4 mg IR-BIC Fasted (N=20) | Fesoterodine 4 mg 10% ER-BIC Fasted (N=20) | Fesoterodine 4 mg 15% ER-BIC Fasted (N=20) | Fesoterodine 4 mg 20% ER-BIC Fasted (N=20) | Fesoterodine 4 mg ER Tablet Fasted (N=20) | Fesoterodine 4 mg 10% ER-BIC Fed (N=20)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Feeling cold (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 1 | 1 | 1 | 0 | 1 | 0
Vessel puncture site pain (General disorders) | 1 | 1 | 1 | 0 | 1 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 1 | 3
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.